CLINICAL TRIAL: NCT03921710
Title: Research Study to Evaluate Capacitation Culture (CAPA) Followed by in Vitro Maturation (IVM) of Human Oocytes: A Randomized Pilot Study
Brief Title: CAPA-IVM Versus STANDARD IVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-2017/QD-CGRH-NCKH&DT
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
  Patients are randomized to either CAPA-IVM or STANDARD-IVM using block randomization by an independent study coordinator using a computer-generated random list (block size 4) on the second day of their periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPA-IVM (Active Comparator): Immature oocytes are culture in the new capacitation-IVM system.
  Interventions: Drug: CAPA-IVM
- Standard-IVM (Active Comparator): Immature oocytes are cultured in the standard IVM system.
  Interventions: Drug: Standard-IVM

INTERVENTIONS:
Drug: CAPA-IVM — Immature oocytes were plated into a 4-well dish (Nunc, Denmark) at 10 COCs/well using CAPA medium (Medicult IVM medium; Origio, Denmark supplemented with 1 mIU/mL rFSH, 5 ng/mL insulin, 10 nM estradiol, 10 mg/mL human serum albumin [SAGE, Denmark] and 25 nM CNP under oil for 24 h at 37°C, 6% carbon dioxide in air). After 24 hours, COCs were washed and transferred into IVM medium (Origio, Denmark) containing 5 ng/mL insulin, 10 nM estradiol, 100 ng/mL human recombinant amphiregulin and 100 mIU/mL rFSH, and incubated under oil for 30 h at 37°C, 6% carbon dioxide in air.
  Arms: CAPA-IVM
Drug: Standard-IVM — Immature oocytes are plated into a 4-well dish at 10 COCs/well using IVM medium supplemented with 75 mIU/mL recombinant FSH (Merck, Switzerland), 100 mIU/mL hCG (MSD, USA), 0.01 mg/mL growth hormone (Merck, Switzerland) and 10 mg/mL human serum albumin (SAGE, Denmark). COCs were incubated for 30 hours at 37°C, 6% carbon dioxide in air.
  Arms: Standard-IVM

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of CAPA-IVM versus standard IVM in women with polycystic ovarian morphology (PCOM) or polycystic ovary syndrome (PCOS) .

DETAILED DESCRIPTION:
Patients preparation

Patients with PCOM are allowed to enroll in the study: (1) women with normal menstrual cycle lengths (≤35 days), and (2) women with oligomenorrhea (menstruation occurring at intervals >35 days with 4-9 periods/year) or total amenorrhea. Patients were followed up until the end of pregnancy.

Patients have their first clinic visit on day 2 of the menstrual cycle. At this visit a blood sample was taken for assessment of FSH (Follicle Stimulating Hormone), LH (Luteinizing Hormone), estradiol and progesterone, and they have their gonadotropin injection 150 IU (international unit) once a day in the afternoon. All patients return in the morning of the next day (cycle day 3) for ultrasound and and the final dose of gonadotropin was given in the afternoon (2pm). When all follicles were <8 mm in diameter, another dose of gonadotropin was given, and patients returned the next day for ultrasound, blood tests and have their final dose of gonadotropin that afternoon (2pm). The maximum number of gonadotropin injections are three, and oocyte retrieval is scheduled at 42-46 hours after the last gonadotropin injection in all patients. Ultrasound and blood tests to determine FSH, LH, estradiol and progesterone levels are performed on the day of OPU (Oocyte Pick-up). During OPU, follicle size is measured before puncture. Larger follicles (≥6 mm) are punctured first, then the needle flushes, then smaller follicles (<6 mm) are punctured. Therefore, each tube contains COCs (Cumulus-Oocyte Complex) of a specific size (<6 or ≥6 mm).

Oocyte culture

Oocytes from patients in the CAPA-IVM group are collected and processed in the presence of CNP (C-type Natriuretic Peptide) as meiotic inhibitor. In the CAPA-IVM group, COCs are plated into a 4-well dish (Nunc, Denmark) at 10 COCs/well using CAPA medium (Medicult IVM medium; Origio, Denmark) supplemented with 1 mIU/mL rFSH, 5 ng/mL insulin, 10 nM estradiol, 10 mg/mL human serum albumin [SAGE, Denmark] and 25 nM (nanoMol) CNP under oil for 24 hours at 37°C, 6% carbon dioxide in air). After 24 hours, COCs are washed and transferred into IVM medium (Origio, Denmark) containing 5 ng/mL insulin, 10 nM estradiol, 100 ng/mL human recombinant amphiregulin and 100 mIU/mL rFSH (recombinant Follicle Stimulating Hormone), and incubated under oil for 30 h at 37°C, 6% carbon dioxide in air.

In the standard IVM group (control), COCs were plated into a 4-well dish at 10 COCs/well using IVM medium supplemented with 75 mIU/mL recombinant FSH (Merck, Switzerland), 100 mIU/mL hCG (MSD, USA), 0.01 mg/mL growth hormone (Merck, Switzerland) and 10 mg/mL human serum albumin (SAGE, Denmark). COCs are incubated for 30 hours using the same physical and atmospheric conditions as the CAPA-IVM group.

Fertilization and embryo culture

After IVM, matured oocytes are fertilized using intracytoplasmic sperm injection (ICSI) and cultured in an incubator at 37°C, 5% carbon dioxide, 5% oxygen. Fertilization check is performed at 16-18 hours after ICSI. Embryos are cultured to day 3 in Global Total LP (Life Global, Canada) in groups of 2-3 embryos per 30 µL microdroplet. Embryos that fulfill the freezing criteria were vitrified (Cryotech, Japan) as cleaving day 3 embryos. Embryos of extremely poor quality (Istanbul consensus on embryo quality assessment) defined as fragmentation >30%, <6 cells, and multi nucleation are not frozen.

Endometrial priming and embryo transfer

No fresh embryo transfers is performed. Patients receive oral estradiol 2 mg 4 times daily from day 2 of their menstrual cycle. After an estradiol treatment period of at least 10 days and when endometrial thickness was ≥8 mm, progesterone 200 mg is administered intra-vaginally 4 times daily. Embryo transfer is scheduled 3 days after starting progesterone. Serum beta hCG is tested 14 days after embryo transfer. If a woman become pregnant, beta human chorionic gonadotropin (hCG) >5 mIU/mL, progesterone administration is maintained at the same dose until at least 11 weeks of pregnancy. An ultrasound scan to determine the viability of pregnancy is performed at 7 weeks' gestation.

Safety of the ART (Assisted Reproductive Technology) procedure in PCOS

Safety is monitored at each clinic visit or, if any side effects occurred, by questioning and examining the patient, with adverse events and serious adverse events recorded on case report forms. Adverse events are defined as any unexpected medical occurrence (symptoms or signs, abnormal laboratory findings or diseases) that emerge or worsen during the trial, relative to the initial trial visit. Possible adverse events including ectopic pregnancy, miscarriage, medication-related reactions such as overdose, sensitivity and toxicity, and any adverse outcomes related to egg collection. Serious adverse events are defined as any unexpected medical occurrence that resulted in death, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacitation. Congenital anomaly or birth defect are considered to be serious adverse events.

Statistical analysis

A key goal of this study is to determine feasibility, acceptability, and outcome variability to aid in planning a larger, adequately-powered efficacy trial. The planned sample size is 80 patients (40 per group), which should allow relatively precise conclusions regarding feasibility outcomes. Given that this is the first time that CAPA-IVM has been used clinically at our center, the objective of this pilot study is to estimate the live birth rate and associated 95% confidence intervals (CI) for the new intervention in clinical practice. Nonparametric statistical methods such as Wilcoxon rank sum is applied to continuous or ordinal outcomes. To estimate 95% confidence intervals (CI) for the difference between two medians, bootstrapping and related resampling methods is applied. The incidence of outcomes is estimated for each treatment group, and the difference between groups was analyzed using relative risk (RR), 95% CI of RR and Fisher exact test. A subgroup analysis is performed based on follicular size (<6 versus ≥6 mm). Data are presented as mean values with standard deviation (SD), medians and interquartile ranges (IQRs), or proportions. All analyses are performed using R (Version 3.0.1; R Foundation for Statistical Computing, Vienna, Austria). Statistical significance is defined as p<0.05.

ELIGIBILITY:
Inclusion criteria:

* < 38 years
* PCOS patients with polycystic ovarian morphology: at least 25 follicles (2-9 mm) throughout the whole ovary and/or increased ovarian volume (>10ml) (it is sufficient that 1 ovary fits these criteria)
* No major uterine or ovarian abnormalities

Exclusion criteria:

* High (>grade 2) grade endometriosis
* Cases with extremely poor sperm (OAT) such as azoospermia or cryptozoospermia

Max Age: 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Wives in infertile couples
Enrollment: 80 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Live birth rate | At least 24 weeks of gestation up to the time of delivery
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twin will be a single count). For the timing of this occur, ongoing pregnancy will be used, i.e. ongoing pregnancy at 12 weeks will be used in calculations, conditional on the fact that this ongoing pregnancy results in live birth.

SECONDARY OUTCOMES:
Ongoing pregnancy rate | At a minimum of 12 weeks from the beginning of the last menstrual cycle
  Pregnancy with detectable heart rate at 12 weeks' gestation
Clinical pregnancy rate | At a minimum of 12 weeks from the beginning of the last menstrual cycle
  Pregnancy with detectable gestational sac at 7 weeks' gestation
Number of oocytes retrieved | Maximum at 30 minutes after oocyte retrieval procedure
  The number of oocyte identified after oocyte retrieval
Oocyte maturation rate | After at least 30 hours of maturation culture
  Rate of mature oocytes on culture oocytes
Number of fertilized oocytes | 16-18 hours after intra-cytoplasmic sperm injection
  Number of fertilized oocyte after sperm insemination
Number of embryos | At least 3 days after intra-cytoplasmic sperm injection
  Number of cleavage embryos obtained
Number of good quality embryos | At least 3 days after intra-cytoplasmic sperm injection
  Number of good cleavage embryos obtained
Number of embryos frozen | At least 3 days after intra-cytoplasmic sperm injection
  Number of cleavage embryos frozen

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — Hope Research Center
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam